CLINICAL TRIAL: NCT01646840
Title: a Phase 1, Open-Label, Single Dose, Relative Bioavailability Study In Healthy Volunteers Comparing PF-04958242 Capsule Formulation To PF-04958242 Oral Solution In The Fasted State
Brief Title: Study Of The PF-04958242 Blood Concentrations Of A Capsule Formulation Of PF-04958242 Compared To A Solution Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1701010
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: PF-04958242; bioequivalence; pharmacokinetics; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — PF-04958242

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04958242 capsule (Experimental)
  Interventions: Drug: PF-04958242 capsule
- PF-04958242 oral solution (Active Comparator)
  Interventions: Drug: PF-04958242 oral solution

INTERVENTIONS:
Drug: PF-04958242 capsule — Single dose of PF-04958242 0.35 mg oral capsule
  Arms: PF-04958242 capsule
Drug: PF-04958242 oral solution — Single dose of PF-04958242 0.35 mg oral solution
  Arms: PF-04958242 oral solution

SUMMARY:
This study will assess the relative bioavailability of a capsule formulation of PF-04958242, relative to a oral solution formulation of PF-04958242 in healthy adult subjects.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (of non childbearing potential) subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Maximum Observed Plasma Concentration (Cmax) | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04958242 | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Plasma Decay Half-Life (t1/2) | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Apparent Oral Clearance (CL/F) | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Apparent Volume of Distribution (Vz/F) | 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 120, and 192 hours post-dose
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | 4 and 192 hours post-dose

SECONDARY OUTCOMES:
no secondary endpoints | no secondary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1701010&StudyName=Study%20Of%20The%20PF-04958242%20Blood%20Concentrations%20Of%20A%20Capsule%20Formulation%20Of%20PF-04958242%20Compared%20To%20A%20Solution%20Formulation